CLINICAL TRIAL: NCT02233634
Title: Impact of Breathing Maneuvers and Oxygen Administration on Myocardial Oxygenation in Patients With Coronary Artery Disease Compared With Healthy Controls - Non-invasive Assessment With Oxygenation-sensitive Cardiovascular Magnetic Resonance Imaging (OS-CMR)
Brief Title: Impact of Breathing Maneuvers on the Oxygenation Supply of the Heart Assessed With MRI in Patients With Coronary Artery Disease
Acronym: CADOS-CMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 107/14; GUDD 1-14 (Other: Inselspital, Institute of Anaesthesiology)
Record Dates: First submitted 2014-09-03; First posted 2014-09-08 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Angiography; Magnetic Resonance Imaging; Oxygen; Hyperoxia; Carbon Dioxide; Apnea; Hyperventilation
MeSH Terms: conditions — Coronary Artery Disease; Hyperoxia; Apnea; Hyperventilation | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAD Patients (Active Comparator): Administration of Oxygen via a mask, Hyperventilation, Combination of Oxygen administration and Hyperventilation, long breath-holds
  Interventions: Drug: Oxygen; Other: Hyperventilation Breath-hold (HVBH); Other: HVBH with Oxygen
- Healthy Volunteers (Control Group) (Active Comparator): Administration of Oxygen via a mask, Hyperventilation, Combination of Oxygen administration and Hyperventilation, long breath-holds
  Interventions: Drug: Oxygen; Other: Hyperventilation Breath-hold (HVBH); Other: HVBH with Oxygen

INTERVENTIONS:
Drug: Oxygen — Oxygen is provided with a standard medical oxygen mask with reservoir (12L/min) for 3-5 min, assigned to both groups
Other: Hyperventilation Breath-hold (HVBH) — 1 Minute of Hyperventilation (25/min) is followed by a consecutive breath-hold for as long as the subject can comfortably tolerate. Both groups will perform this maneuver
Other: HVBH with Oxygen — 1 Minute of Hyperventilation (25/min) with an oxygen mask mounted (12L/min) is followed by a consecutive breath-hold for as long as the subject can comfortably tolerate. Both groups will perform this maneuver

SUMMARY:
Patients with an impaired blood supply of the heart routinely receive oxygen in order to improve or preserve the oxygen supply of the heart muscle in acute cardiac care. In recent studies a new innovative MRI-technique that can detect changes in oxygen supply of the heart was able to show that the administration of oxygen or fast breathing can decrease the blood supply of the arteries supplying the heart muscle with oxygen. Thus, the administration of oxygen may paradoxically impair the oxygen supply of the heart muscle. In this study the investigators want to investigate, whether the administration of exogenous oxygen via a mask alone and in combination with fast breathing leads to a decrease in oxygen supply in regions with already impaired blood supply by a narrowing of a coronary artery of the heart.

DETAILED DESCRIPTION:
Background

Patients with acute myocardial ischemia receive oxygen as a standard measure of care to maintain or improve the myocardial oxygen supply. In 1975 Neil et al. were able to show that higher oxygen concentration reduces myocardial blood flow. However, since the oxygen concentration in the blood was significantly increased it was/is assumed that the higher oxygen supply outweighs the decrease in perfusion. Oxygenation-Sensitive (OS) Cardiovascular Magnetic Resonance (CMR) is a newer technology that uses the paramagnetic deoxyhemoglobin in the blood as an endogenous contrast. An drop in tissue oxygenation (drop in oxyhemoglobin) results in an increase in deoxyhemoglobin, which results in an drop in SI in OS-images. Vice versa an increase in tissue oxygenation results in an increase in OS-SI. Therefore, OS-CMR can assess myocardial tissue oxygenation changes non-invasively, free of contrast and free of radiation. While other diagnostic modalities only give information on myocardial oxygenation with surrogate parameters that may indicate ischemia OS-CMR gives local functional information of the myocardial oxygen supply. Studies have been performed using OS-CMR for the detection of coronary artery disease. More recently breathing maneuvers that change systemic blood gases have been suggested as a vasoactive stimulus to detect coronary artery disease and measure changes to the myocardial oxygen supply. Guensch et al. were able to show that hypercapnia and the combination of hypercapnia and hypoxia lead to a increase of myocardial oxygenation that can only be explained by an increase blood flow. However, hypocapnia resulted in a decrease in myocardial oxygenation in healthy volunteers. In a porcine model the investigators were able to show that the increase in systemic oxygen supply resulted in a decrease in myocardial blood flow in healthy and swine with an acute coronary artery stenosis, but a decrease in myocardial oxygenation was only observed in the animals with a coronary artery stenosis (Abstract Guensch et al: Administration of exogenous oxygen may worsen myocardial ischemia, ESC 2014, accepted). The impact of hyperoxia as well as hypocapnia and hypercapnia in humans with a chronic coronary artery disease is poorly investigated. As the administration of oxygen is part of the treating guidelines in acute myocardial ischemia and in certain situations (e.g. anesthesia) higher oxygen concentrations are maintained for safety reasons, it is important to further investigate the role of higher oxygen concentrations in coronary artery disease. Further the investigators want to shed light on transient states of hypocapnia and hypercapnia induced by voluntary breathing. Because OS-CMR is a safe diagnostic tool (no radiation, no contrast, no pharmacologic vasodilator required) and can give insight on the oxygenation changes of the heart is it ideal to test the hypothesis. Therefore the investigators want to invite patients with a known coronary stenosis (confirmed by previous coronary angiography) scheduled for a percutaneous coronary intervention (staged PCI) or coronary artery bypass surgery to participate in this study prior to the intervention and compare the MRI results to healthy volunteers. All participants will perform hyperventilation with a consecutive breath-hold as well as inhale oxygen for 3-5 minutes while the breathing maneuver is being repeated. For the patients the results will then be compared to the findings of coronary angiography (QCA, reduction in lumen-diameter of the vessel).

Objective

With this study the investigators want to investigate whether the administration of oxygen, as well as performing breathing maneuvers (hyperventilation, breath-holding) have a negative or positive effect on the oxygenation of myocardium subtended to arteries diseased of coronary artery disease, as opposed to healthy subjects.

Methods

CAD-patients with a known coronary pathology that are scheduled for a PCI or coronary bypass surgery will be recruited for the CMR exam prior to the coronary intervention. A i.v. line will be placed for safety reason. During short breath-holds oxygenation-sensitive baseline images and cardiac function images will be acquired. The subjects will then be asked to hyperventilate for one minute with 20-30 breaths/min. Immediately after a maximal breath-hold will be performed in end-expiration as long as the subject can comfortably bear. During the entire breath-hold oxygenation sensitive images will be recorded. Whenever the subject feels the need to breath, he/she can immediately do so and signal the technician with a call bell. After recovery the subject will breath oxygen 12-15L/min through a mask for 3-5 min after which oxygenation sensitive images as well as function images will be repeated. The hyperventilation-breath-hold will be repeated with oxygen. Healthy volunteers will undergo the same protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known relevant coronary artery stenosis (defined by previous coronary angiography, QCA: reduction in lumen-diameter of the vessel >50%) with a scheduled intervention or operation to treat this stenosis (staged PCI or coronary artery bypass surgery)
* CMR feasible prior to intervention or surgery
* Age ≥18 years
* Written informed consent
* For healthy participants: Absence of cardiovascular and lung disease, and absence of medication with cardiovascular effects
* Absence of exclusion criteria

Exclusion Criteria

* General Contraindication against MRI-Scans: (claustrophobia, ferromagnetic implants, clips, pacemakers, shrapnels, ophthalmic metal deposits)
* Pregnancy or inconclusive test result
* Age <18 years
* Inability to give informed consent
* Consumption of caffeine, tea, treatment of dipyridamol <12h before the scan
* Medication with calcium antagonists (ok, if can be paused on the day of the scan)
* Constant medication with nitrates (ok, if can be paused on the day of the scan)
* Medication with methyl-xanthines
* Acute myocardial ischemia/myocardial infarction
* Previous Coronary Bypass Surgery
* Pulmonary Disease
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Presence of cardiac or lung disease for healthy volunteers, nicotine consumption within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Change of signal intensity (SI) in oxygenation-sensitive (OS) Cardiovascular Magnetic Resonance (CMR) during the breathing maneuvers/oxygen administration | During CMR scan, expected to be on average approx. 45 minutes

SECONDARY OUTCOMES:
Comparison of OS-SI changes between healthy and post-stenotic myocardium during the breathing-maneuvers/oxygen administration in CAD patients | During CMR scan, expected to be on average approx. 45 minutes
Comparison of OS-SI changes between healthy volunteers and and CAD patients during the breathing-maneuvers/oxygen administration | During CMR scan, expected to be on average approx. 45 minutes
Comparison between OS-SI changes during the breathing maneuvers/oxygen administration and results in quantitative coronary angiography in CAD patients (reduction of lumen diameter) | During CMR scan, expected to be on average approx. 45 minutes, and the subsequent coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Balthasar Eberle, MD, Principal Investigator — Department of Anaesthesiology and Pain Therapy, Bern University Hospital, Inselspital, Bern
Locations (1):
- Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Guensch DP, Fischer K, Flewitt JA, Friedrich MG. Impact of intermittent apnea on myocardial tissue oxygenation--a study using oxygenation-sensitive cardiovascular magnetic resonance. PLoS One. 2013;8(1):e53282. doi: 10.1371/journal.pone.0053282. Epub 2013 Jan 3. PMID 23301055
- [Background] Guensch DP, Fischer K, Flewitt JA, Yu J, Lukic R, Friedrich JA, Friedrich MG. Breathing manoeuvre-dependent changes in myocardial oxygenation in healthy humans. Eur Heart J Cardiovasc Imaging. 2014 Apr;15(4):409-14. doi: 10.1093/ehjci/jet171. Epub 2013 Sep 27. PMID 24078154
- [Background] Guensch DP, Fischer K, Flewitt JA, Friedrich MG. Myocardial oxygenation is maintained during hypoxia when combined with apnea - a cardiovascular MR study. Physiol Rep. 2013 Oct;1(5):e00098. doi: 10.1002/phy2.98. Epub 2013 Oct 11. PMID 24303170
- [Background] Luu JM, Friedrich MG, Harker J, Dwyer N, Guensch D, Mikami Y, Faris P, Hare JL. Relationship of vasodilator-induced changes in myocardial oxygenation with the severity of coronary artery stenosis: a study using oxygenation-sensitive cardiovascular magnetic resonance. Eur Heart J Cardiovasc Imaging. 2014 Dec;15(12):1358-67. doi: 10.1093/ehjci/jeu138. Epub 2014 Aug 7. PMID 25104812
- [Background] Neill WA, Hattenhauer M. Impairment of myocardial O2 supply due to hyperventilation. Circulation. 1975 Nov;52(5):854-8. doi: 10.1161/01.cir.52.5.854. PMID 1175266
- [Background] Momen A, Mascarenhas V, Gahremanpour A, Gao Z, Moradkhan R, Kunselman A, Boehmer JP, Sinoway LI, Leuenberger UA. Coronary blood flow responses to physiological stress in humans. Am J Physiol Heart Circ Physiol. 2009 Mar;296(3):H854-61. doi: 10.1152/ajpheart.01075.2007. Epub 2009 Jan 23. PMID 19168724
- [Background] Nakao K, Ohgushi M, Yoshimura M, Morooka K, Okumura K, Ogawa H, Kugiyama K, Oike Y, Fujimoto K, Yasue H. Hyperventilation as a specific test for diagnosis of coronary artery spasm. Am J Cardiol. 1997 Sep 1;80(5):545-9. doi: 10.1016/s0002-9149(97)00419-0. PMID 9294979
- [Derived] Guensch DP, Fischer K, Yamaji K, Luescher S, Ueki Y, Jung B, Erdoes G, Grani C, von Tengg-Kobligk H, Raber L, Eberle B. Effect of Hyperoxia on Myocardial Oxygenation and Function in Patients With Stable Multivessel Coronary Artery Disease. J Am Heart Assoc. 2020 Mar 3;9(5):e014739. doi: 10.1161/JAHA.119.014739. Epub 2020 Feb 22. PMID 32089047
- [Derived] Fischer K, Yamaji K, Luescher S, Ueki Y, Jung B, von Tengg-Kobligk H, Windecker S, Friedrich MG, Eberle B, Guensch DP. Feasibility of cardiovascular magnetic resonance to detect oxygenation deficits in patients with multi-vessel coronary artery disease triggered by breathing maneuvers. J Cardiovasc Magn Reson. 2018 May 7;20(1):31. doi: 10.1186/s12968-018-0446-y. PMID 29730991
- See also: Explanation and Study Results of a Hyperventilation Breath-Hold in Healthy Volunteers as used in the protocol — http://www.jcmr-online.com/content/16/S1/P49